CLINICAL TRIAL: NCT02848495
Title: Genetic Study on the Familial Forms of Intracranial Aneurysm
Brief Title: Biocollection on the Familial Forms of Intracranial Aneurysm
Acronym: GAÏA
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC12_0458
Record Dates: First submitted 2016-07-21; First posted 2016-07-28 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Intracranial Aneurysm
Keywords: Aneurysm; Biocollection; Familial Form
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For one patient included: Ethylenediaminetetraacetic acid (EDTA) tubes for DNA (20 mL blood)
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: Non-Interventional

SUMMARY:
Intracranial aneurysm (IA) is an asymptomatic cerebrovascular abnormality affecting 3.2% of the general population. The devastating complication of IA is its rupture, resulting in subarachnoid haemorrhage that can lead to severe disability and death.

Unfortunately, there are neither reliable clues nor diagnostic tools to predict the formation and/or the fate of an IA in a given individual. Also, there is no pharmacological drug available to prevent the rupture of aneurysm and subsequent subarachnoid haemorrhage. Current treatments are invasive with a significant risk of procedural morbidity. Thus, still now, the management of patients with IA remains extremely challenging and still controversial.

Although the pathogenesis of IA has been the subject of many studies for the last decade, the mechanisms underlying IA formation, growth and rupture are still mostly unknown and relevant animal models of IA are not available.

Familial history of IA predisposes to IA formation and rupture and increasing evidence suggest a genetic component of IA formation, with heterogeneous modes of inheritance and penetrance.

This project, gathering neuroradiologists, geneticists and vascular biologists, addresses the urgent need to understand the pathogenic mechanisms of IA to develop diagnostic and predictive tools of risk of IA.

The investigators propose to identify IA-causing variants by whole-exome sequencing in familial forms of the disease.

The investigators hypothesises that the functional analysis of the causal / susceptibility variants thus identified will provide clues to understanding the pathological mechanisms of IA formation, and the bases for developing diagnostic tools. This project aims at meeting this challenge. Based on preliminary data that already allowed to identify such a variant, and the combination of genetic and functional investigations, the specific objectives of this project are: - To identify IA-causing variants in familial forms of the disease by whole-exome sequencing; - To understand the function of these genes/ variants in the formation and rupture of IA by molecular and cellular approaches and generation of relevant animal models; - To discover potential biomarkers of risk of IA formation and/or rupture.

ELIGIBILITY:
Inclusion criteria :

* Inclusion criteria indexes and related cases (familial) of intracranial aneurysms:

  * Index: Any patient consulting for a major IA and some typical bifurcation with at least one other case reached akin IA 1st degree
  * Related: All similar to the first degree, aged 20 or more, patients with a family background of IA and some typical bifurcation (≥2 achieved) For the latter, directed by screening with Magnetic resonance imaging (MRI) sequence Time of Flight (TOF), axial T2, EGT2.
  * Consent oral and in writing to the Biocollection consent Form for participation in the collection of biological samples
* Inclusion criteria sporadic cases of IA:

  * Any patient consulting for IA and some typical bifurcation
  * Patients aged of 20 years or older
  * Consent oral and in writing to the Biocollection consent Form for participation in the collection of biological samples

Exclusion Criteria :

- Non Inclusion Criteria:

* Patients who have shown the inability or have refused to sign the consent informed biocollection
* Syndromic diagnosis known as IA provider
* Marfan Syndrome
* AOS with SMAD 3
* Danlos Syndrome Elhers type II and IV
* Autosomal Dominant Polycystic
* Moyamoya Syndrome
* Character of IA:
* Dissecting or fusiform
* Combined with an arteriovenous malformation
* Blister-like
* Mycotic
* Pathology of the cerebral white matter detected on MRI, evoking:
* COL4A1 mutation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The initial stage of this biocollection based on the recruitment of large families for genetic linkage analysis.
  In the first instance, we identify patients with intracranial aneurysms occurring in a family context, and to conduct a comprehensive investigation according to clinical guidelines in force to assess the potentially informative family and ensure their adherence to the prior biocollection. The next step consists on the fine and accurate phenotyping of each of the family members (imaging) and the collection of a blood sample for DNA extraction for molecular genetic analysis.
  The population recruited will be composed of index and their healthy relatives and cases with sporadic cases and IA. The kinship links will be established from family trees.
Sampling Method: Non-Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
DNA analysis to identify new genes (and new physiological pathways) associated to the risk of intracranial aneurysm | Until one year

CONTACTS AND LOCATIONS:
Overall Officials: Romain BOURCIER, PhD, Principal Investigator — Nantes University Hospital
Locations (8):
- France (8):
  - AP-HP, Henri Mondor hospital, Créteil
  - CHD La Roche sur YON, La Roche-sur-Yon
  - Nantes University Hospital, Nantes
  - University Hospital Poitiers, Poitiers
  - University Hospital Rennes, Rennes
  - Rouen University Hospital, Rouen
  - Bordeaux University Hospital, Talence
  - Tours University Hospital, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canham PB, Finlay HM. Morphometry of medial gaps of human brain artery branches. Stroke. 2004 May;35(5):1153-7. doi: 10.1161/01.STR.0000124926.76836.df. Epub 2004 Mar 11. PMID 15017007
- [Background] Rhoton AL Jr. Aneurysms. Neurosurgery. 2002 Oct;51(4 Suppl):S121-58. No abstract available. PMID 12234448
- [Background] Rinkel GJ, Djibuti M, Algra A, van Gijn J. Prevalence and risk of rupture of intracranial aneurysms: a systematic review. Stroke. 1998 Jan;29(1):251-6. doi: 10.1161/01.str.29.1.251. PMID 9445359
- [Background] Vlak MH, Algra A, Brandenburg R, Rinkel GJ. Prevalence of unruptured intracranial aneurysms, with emphasis on sex, age, comorbidity, country, and time period: a systematic review and meta-analysis. Lancet Neurol. 2011 Jul;10(7):626-36. doi: 10.1016/S1474-4422(11)70109-0. PMID 21641282
- [Background] Ronkainen A, Hernesniemi J, Ryynanen M. Familial subarachnoid hemorrhage in east Finland, 1977-1990. Neurosurgery. 1993 Nov;33(5):787-96; discussion 796-97. doi: 10.1227/00006123-199311000-00001. PMID 8264874
- [Derived] Haemmerli J, Morel S, Georges M, Haidar F, Chebib FT, Morita A, Nozaki K, Tominaga T, Bervitskiy AV, Rzaev J, Schaller K, Bijlenga P. Characteristics and Distribution of Intracranial Aneurysms in Patients with Autosomal Dominant Polycystic Kidney Disease Compared with the General Population: A Meta-Analysis. Kidney360. 2023 Apr 1;4(4):e466-e475. doi: 10.34067/KID.0000000000000092. Epub 2023 Feb 20. PMID 36961086
- [Derived] Zuurbier CCM, Bourcier R, Constant Dit Beaufils P, Redon R, Desal H; ICAN Investigators; Bor ASE, Rinkel GJE, Greving JP, Ruigrok YM. Risk Prediction of New Intracranial Aneurysms at Follow-Up Screening in People With a Positive Family History. Stroke. 2023 Apr;54(4):1015-1020. doi: 10.1161/STROKEAHA.122.041393. Epub 2023 Feb 27. PMID 36846982
- [Derived] Zuurbier CCM, Bourcier R, Constant Dit Beaufils P, Redon R, Desal H; ICAN Investigators; Bor ASE, Lindgren AE, Rinkel GJE, Greving JP, Ruigrok YM. Number of Affected Relatives, Age, Smoking, and Hypertension Prediction Score for Intracranial Aneurysms in Persons With a Family History for Subarachnoid Hemorrhage. Stroke. 2022 May;53(5):1645-1650. doi: 10.1161/STROKEAHA.121.034612. Epub 2022 Feb 11. PMID 35144487
- [Derived] Bakker MK, van der Spek RAA, van Rheenen W, Morel S, Bourcier R, Hostettler IC, Alg VS, van Eijk KR, Koido M, Akiyama M, Terao C, Matsuda K, Walters RG, Lin K, Li L, Millwood IY, Chen Z, Rouleau GA, Zhou S, Rannikmae K, Sudlow CLM, Houlden H, van den Berg LH, Dina C, Naggara O, Gentric JC, Shotar E, Eugene F, Desal H, Winsvold BS, Borte S, Johnsen MB, Brumpton BM, Sandvei MS, Willer CJ, Hveem K, Zwart JA, Verschuren WMM, Friedrich CM, Hirsch S, Schilling S, Dauvillier J, Martin O; HUNT All-In Stroke; China Kadoorie Biobank Collaborative Group; BioBank Japan Project Consortium; ICAN Study Group; CADISP Group; Genetics and Observational Subarachnoid Haemorrhage (GOSH) Study investigators; International Stroke Genetics Consortium (ISGC); Jones GT, Bown MJ, Ko NU, Kim H, Coleman JRI, Breen G, Zaroff JG, Klijn CJM, Malik R, Dichgans M, Sargurupremraj M, Tatlisumak T, Amouyel P, Debette S, Rinkel GJE, Worrall BB, Pera J, Slowik A, Gaal-Paavola EI, Niemela M, Jaaskelainen JE, von Und Zu Fraunberg M, Lindgren A, Broderick JP, Werring DJ, Woo D, Redon R, Bijlenga P, Kamatani Y, Veldink JH, Ruigrok YM. Genome-wide association study of intracranial aneurysms identifies 17 risk loci and genetic overlap with clinical risk factors. Nat Genet. 2020 Dec;52(12):1303-1313. doi: 10.1038/s41588-020-00725-7. Epub 2020 Nov 16. PMID 33199917
- [Derived] Bourcier R, Le Scouarnec S, Bonnaud S, Karakachoff M, Bourcereau E, Heurtebise-Chretien S, Menguy C, Dina C, Simonet F, Moles A, Lenoble C, Lindenbaum P, Chatel S, Isidor B, Genin E, Deleuze JF, Schott JJ, Le Marec H; ICAN Study Group; Loirand G, Desal H, Redon R. Rare Coding Variants in ANGPTL6 Are Associated with Familial Forms of Intracranial Aneurysm. Am J Hum Genet. 2018 Jan 4;102(1):133-141. doi: 10.1016/j.ajhg.2017.12.006. PMID 29304371